CLINICAL TRIAL: NCT06908694
Title: GLP1-Receptor Agonists in Men With Prostate Cancer: Control of Cardiovascular Risk Factors and Prostate Biomarkers
Brief Title: Investigation of GLP1-Receptor Agonists in Men With Prostate Cancer Taking Androgen Deprivation Therapy
Acronym: GAINPCCONTROL
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5100
Record Dates: First submitted 2025-03-26; First posted 2025-04-03 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-03

CONDITIONS: Prostate Cancer
Keywords: Androgen Deprivation Therapy; GLP-1 Receptor Agonists
MeSH Terms: conditions — Prostatic Neoplasms | interventions — semaglutide

STUDY DESIGN:
Intervention Model Description: Open-label single-arm phase IV trial.
  Following enrolment, all participants will undergo a baseline visit, a 1-month telephone follow-up visit, 3-month visit, 6-month and 12-month (Close-out) visit.
  The semaglutide dose will be 0.25mg subcutaneously once weekly for weeks 1-4, then 0.5mg once weekly for weeks 5-8, then 1mg once weekly for weeks 9-12, then 1.7mg once weekly for weeks 13-16, and then 2.4mg for the remainder of the trial. Semaglutide dose may be decreased in the case of adverse events to the highest tolerated dose.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Semaglutide (Experimental): The semaglutide dose will be 0.25mg subcutaneously once weekly for weeks 1-4, then 0.5mg once weekly for weeks 5-8, then 1mg once weekly for weeks 9-12, then 1.7mg once weekly for weeks 13-16, and then 2.4mg for the remainder of the trial. Semaglutide dose may be decreased in the case of adverse events to the highest tolerated dose.
  Interventions: Drug: Semaglutide Pen Injector

INTERVENTIONS:
Drug: Semaglutide Pen Injector — The semaglutide dose will be 0.25mg subcutaneously once weekly for weeks 1-4, then 0.5mg once weekly for weeks 5-8, then 1mg once weekly for weeks 9-12, then 1.7mg once weekly for weeks 13-16, and then 2.4mg for the remainder of the trial. Semaglutide dose may be decreased in the case of adverse events to the highest tolerated dose.
  Other Names: Wegovy®

SUMMARY:
GAIN PC CONTROL is a study investigating Glucagon-Like Peptide-1 Receptor Agonists in men with prostate cancer who are being treated with androgen deprivation therapy.

DETAILED DESCRIPTION:
GAIN PC CONTROL is an open-label single-arm phase IV trial that will evaluate 1) the safety and tolerability of Glucagon-Like Peptide-1 Receptor Agonists (GLP-1 RAs) in men with prostate cancer (PC) treated with androgen deprivation therapy (ADT); 2) the effects of GLP-1 RAs on weight, waist circumference, blood pressure, HbA1c, lipids, PSA and Creatinine, estimated glomerular filtration rate in men with PC treated with ADT.

Patients who meet eligibility criteria and who provide informed consent will be enrolled to receive semaglutide.

Following enrollment, all participants will undergo a baseline visit, a 1-month telephone follow-up visit, 3-month visit, 6-month and a 12-month (Close-out) visit.

The semaglutide dose will be 0.25mg subcutaneously once weekly for weeks 1-4, then 0.5mg once weekly for weeks 5-8, then 1mg once weekly for weeks 9-12, then 1.7mg once weekly for weeks 13-16, and then 2.4mg for the remainder of the trial. Semaglutide dose may be decreased in the case of adverse events to the highest tolerated dose.

ELIGIBILITY:
Inclusion Criteria:

* Have a physician diagnosis of PC
* Must be receiving or planned to receive ADT (gonadotropin releasing hormone agonist or antagonist ± androgen receptor pathway inhibitor)
* Elevated BMI

  1. ≥30kg/m2 or
  2. ≥27kg/m2 in the presence of at least one of hypertension, type 2 diabetes, obstructive sleep apnea or dyslipidemia

Exclusion Criteria:

* Type 1 diabetes
* Taking a GLP-1 RA
* <18 years of age
* History of pancreatitis
* Personal or family history of medullary cancer of the thyroid
* Multiple endocrine neoplasia type 2

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of Serious Adverse Events | 12 months
  An event that leads to death; is life-threatening; results in hospitalization or its prolongation; disability or permanent damage; congenital anomaly or birth defect; or other medical event that is considered serious.
Number of Adverse Events leading to Drug Discontinuation | 6 months
  Adverse Events leading to Drug Discontinuation
Measure of Weight | 12 months
  Measure of Weight
Measure of Waist Circumference | 12 months
  Measure of Waist Circumference
Measure of Blood Pressure | 12 months
  Measure of Blood Pressure
Concentration of HbA1c | 12 months
  Concentration of HbA1c
Concentration of Lipids | 12 months
  Total Cholesterol, low-density lipoprotein cholesterol, high-density lipoprotein cholesterol, triglycerides
Concentration of PSA | 12 months
  Concentration of PSA
Concentration of Creatinine | 12 months
  Concentration of Creatinine
Calculation of estimated glomerular rate | 12 months
  Calculation of estimated glomerular rate
Number of Clinical Outcomes | 12 months
  Death, Hospitalization, New Diabetes, Myocardial Infarction, Stroke, Heart Failure, Peripheral Arterial Disease, Venous Thromboembolism

CONTACTS AND LOCATIONS:
Overall Officials: Darryl Leong, MBBs,MPH,PhD,FRACP,FESC, Principal Investigator — Population Health Research Institute and McMaster University; Jehonathan Pinthus, MD,FRCS(C),PhD, Principal Investigator — Juravinski Cancer Centre
Locations (1):
- Juravinski Cancer Centre, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No